CLINICAL TRIAL: NCT04105660
Title: Recovery From Propofol Anaesthesia Guided by Frontal EEG Wave Analysis Compared to Bispectral Index Monitoring Alone in Laparoscopic Surgery: A Multicentre Double-blind Randomised Controlled Trial
Brief Title: Electroencephalogram (EEG) in General Anaesthesia - More Than Only a Bispectral Index (BIS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Cantonal Hospital of Graubünden, Chur, Switzerland (Unknown); University Hospital, Geneva (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2019-00132
Record Dates: First submitted 2019-09-17; First posted 2019-09-26 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Anesthesia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): EEG monitoring in addition to standard monitoring (clinical parameters and BIS index)
  Interventions: Other: Training for EEG monitoring; Other: Standard monitoring
- Control arm (Active Comparator): Standard monitoring including clinical parameters and BIS index
  Interventions: Other: Standard monitoring

INTERVENTIONS:
Other: Training for EEG monitoring — Training for reading EEG curves during anaesthesia
  Arms: Intervention arm
Other: Standard monitoring — Standard monitoring including clinical parameters and BIS index

SUMMARY:
Processed electroencephalogram (EEG) monitors are routinely used in addition to clinical parameters to assess the depth of anaesthesia during general anaesthesia.

DETAILED DESCRIPTION:
Processed electroencephalogram (EEG) monitors are routinely used in addition to clinical parameters to assess the depth of anaesthesia during general anaesthesia. In addition to the bispectral (BIS) index displayed as an index, the raw frontal EEG can be displayed as a curve on these monitors. After a short training, anaesthetists might be more accurate and faster in assessing depth of anaesthesia by recognizing the pattern of the EEG curve than by using the BIS index. This may further enhance the positive effects that could be demonstrated for the use of BIS monitors.

Therefore, the aim of the investigator's study is to investigate the clinical relevance of interpreting the raw frontal EEG in addition to only using the BIS index for titrating intravenous anaesthetics.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing in-hospital laparoscopic abdominal surgery with general anaesthesia using Propofol based on the Schnider model (target controlled infusion)42, 43
* Minimal duration of surgery of 60 minutes
* Written informed consent

Exclusion Criteria:

* Same-day surgery
* Language barrier
* Patients under 18 years of age
* Pregnancy (using a beta-human chorionic gonadotropin (HCG) measurement in a blood sample of women in childbearing age)
* Allergy to Propofol
* Administration of hypnotics other than Propofol, such as ketamine or midazolam preoperatively or intraoperatively
* Known brain pathology, such as seizure disorders, dementia, cerebrovascular disease or brain death

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-05-28 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Quality of recovery (QoR): QoR-15 scale | 24 hours after surgery
  QoR-15 scale (scale from 0 to 150; 0 means best, 150 worst recovery)

SECONDARY OUTCOMES:
Propofol consumption | during anaesthesia
  Propofol consumption in mg/kg/h
Quality of recovery (QoR): QoR-15 scale | 48 hours after surgery
  QoR-15 scale (scale from 0 to 150; 0 means best, 150 worst recovery)
Time spent in postanaesthesia care unit (PACU) | At arrival to and at discharge from postanaesthesia care unit (an average of 120 minutes)
  Time in minutes from arrival in PACU until discharge from PACU
Time to extubation | At time of skin closure and at time of extubation (an average of 90 minutes)
  Time in minutes from skin closure to extubation
Risk of awareness | daily from admission up to hospital discharge, an average of approximately 14 days
  Brice interview daily until hospital discharge
Aldrete score | Once at discharge from postanaesthesia care unit (PACU), approximately on day 2 of admission to hospital
  Measurement of recovery; score is 0 to 10, 0 means worst recovery, 10 means best recovery
Incidence of Postoperative Nausea and Vomiting (PONV) | daily from admission up to hospital discharge, an average of approximately 14 days
  Incidence of nausea and vomiting daily until hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Salome Dell-Kuster, MD MSc, Principal Investigator — University Hospital, Basel, Switzerland; Christoph S Burkhart, MD, Principal Investigator — Cantonal Hospital Graubünden
Locations (4):
- Switzerland (4):
  - Cantonal Hospital Aarau, Aarau
  - University Hospital Basel, Basel
  - Cantonal Hospital Graubünden, Chur
  - Clinic of Anaesthesiology, Geneva

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data will be available upon reasonable request from the last authors of this publication (Christoph S. Burkhart, ORCID 0000-0002-9288-117X and Salome Dell-Kuster, ORCID 0000-0001-7219-7138)

REFERENCES:
- [Derived] Gruber BU, Girsberger V, Kusstatscher L, Funk S, Luethy A, Jakus L, Maillard J, Steiner LA, Dell-Kuster S, Burkhart CS. Comparing propofol anaesthesia guided by Bispectral Index monitoring and frontal EEG wave analysis with standard monitoring in laparoscopic surgery: protocol for the 'EEG in General Anaesthesia - More Than Only a Bispectral Index' Trial, a multicentre, double-blind, randomised controlled trial. BMJ Open. 2022 Jun 10;12(6):e059919. doi: 10.1136/bmjopen-2021-059919. PMID 35688587